CLINICAL TRIAL: NCT02046512
Title: Randomized Controlled Trial of Lactobacillus Rhamnosus GG to Promote Intestinal Health
Brief Title: Probiotics to Promote Intestinal Health
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201310102; CK000162-aim3 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Communicable Diseases; Infection; Anti-Infective Agents; Therapeutic Uses; Pharmacologic Actions
Keywords: Probiotics
MeSH Terms: conditions — Communicable Diseases; Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Patients randomized to probiotic therapy will receive 1 capsule containing 10 billion cells of Lactobacillus rhamnosus GG on a twice-daily basis
  Interventions: Dietary Supplement: Probiotic
- Sugar Pill (Placebo Comparator): Patients randomized to placebo therapy will receive an identical appearing placebo capsule on a twice-daily basis
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — 1 capsule containing 10 billion cells of Lactobacillus rhamnosus GG on a twice-daily basis
  Other Names: Culturelle
  Arms: Probiotic
Other: Placebo — Sugar pill
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to evaluate the effectiveness of bacteria called Lactobacillus GG, a Probiotic, in preventing the growth of resistant bacteria in the digestive tract in patients on broad spectrum antimicrobials.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old
* Admission to the non-ICU medical and surgical wards
* On broad spectrum antimicrobials with an anticipated length of stay of >48 hours

Exclusion Criteria:

* Pregnancy
* Non English speaking
* Expected to die within 7 days
* Unable or unwilling to consent
* HIV infection with a CD4 count <200
* Neutropenia with an absolute neutrophil count less than 500 cells/ml (or expected to drop to less than 500)
* Clinically significant diarrhea or history of C. difficile infection in the last 3 months
* History of VRE colonization and/or infection in the last year
* Transplant recipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Lucado J, Gould C, Elixhauser A. Clostridium Difficile Infections (CDI) in Hospital Stays, 2009. 2012 Jan. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #124. Available from http://www.ncbi.nlm.nih.gov/books/NBK92613/ PMID 22574332
- [Background] Hall AJ, Curns AT, McDonald LC, Parashar UD, Lopman BA. The roles of Clostridium difficile and norovirus among gastroenteritis-associated deaths in the United States, 1999-2007. Clin Infect Dis. 2012 Jul;55(2):216-23. doi: 10.1093/cid/cis386. Epub 2012 Apr 4. PMID 22491338
- [Background] Yahav D, Lador A, Paul M, Leibovici L. Efficacy and safety of tigecycline: a systematic review and meta-analysis. J Antimicrob Chemother. 2011 Sep;66(9):1963-71. doi: 10.1093/jac/dkr242. Epub 2011 Jun 18. PMID 21685488
- [Background] Kelesidis T, Humphries R, Uslan DZ, Pegues DA. Daptomycin nonsusceptible enterococci: an emerging challenge for clinicians. Clin Infect Dis. 2011 Jan 15;52(2):228-34. doi: 10.1093/cid/ciq113. PMID 21288849
- [Background] Infectious Diseases Society of America (IDSA); Spellberg B, Blaser M, Guidos RJ, Boucher HW, Bradley JS, Eisenstein BI, Gerding D, Lynfield R, Reller LB, Rex J, Schwartz D, Septimus E, Tenover FC, Gilbert DN. Combating antimicrobial resistance: policy recommendations to save lives. Clin Infect Dis. 2011 May;52 Suppl 5(Suppl 5):S397-428. doi: 10.1093/cid/cir153. No abstract available. PMID 21474585
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: carbapenem-resistant Enterobacteriaceae. MMWR Morb Mortal Wkly Rep. 2013 Mar 8;62(9):165-70. PMID 23466435
- [Background] Morrow LE, Kollef MH, Casale TB. Probiotic prophylaxis of ventilator-associated pneumonia: a blinded, randomized, controlled trial. Am J Respir Crit Care Med. 2010 Oct 15;182(8):1058-64. doi: 10.1164/rccm.200912-1853OC. Epub 2010 Jun 3. PMID 20522788
- [Background] Goldenberg JZ, Ma SS, Saxton JD, Martzen MR, Vandvik PO, Thorlund K, Guyatt GH, Johnston BC. Probiotics for the prevention of Clostridium difficile-associated diarrhea in adults and children. Cochrane Database Syst Rev. 2013 May 31;(5):CD006095. doi: 10.1002/14651858.CD006095.pub3. PMID 23728658
- [Background] Johnston BC, Ma SS, Goldenberg JZ, Thorlund K, Vandvik PO, Loeb M, Guyatt GH. Probiotics for the prevention of Clostridium difficile-associated diarrhea: a systematic review and meta-analysis. Ann Intern Med. 2012 Dec 18;157(12):878-88. doi: 10.7326/0003-4819-157-12-201212180-00563. PMID 23362517
- [Background] Hink T, Burnham CA, Dubberke ER. A systematic evaluation of methods to optimize culture-based recovery of Clostridium difficile from stool specimens. Anaerobe. 2013 Feb;19:39-43. doi: 10.1016/j.anaerobe.2012.12.001. Epub 2012 Dec 13. PMID 23247066

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Probiotic | Sugar Pill
Started | 45 | 44
Completed | 44 | 44
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotic | Sugar Pill | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Customized [Median (Full Range); unit: years]
  Age | 58 [25 to 92] | 60 [23 to 81] | 59 [23 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 22 | 24 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 25 | 49
  Non-white | 20 | 19 | 39
Region of Enrollment [Number; unit: participants]
  United States | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acquisition of Any New Antibiotic-resistant Organism
Description: Acquisition in the gastrointestinal tract of any new antibiotic resistant organism post-enrollment. Antibiotic resistant organisms include: C. difficile, vancomycin-resistant enterococci (VRE), multidrug-resistant Acinetobacter baumannii, multidrug-resistant Pseudomonas, ciprofloxacin-resistant Enterobacteriaceae, extended-spectrum betalactamase (ESBL) producing Enterobacteriaceae.
Time Frame: Outcome will be measured approximately every 3 days after enrollment throughout hospitalization, and at the time of discharge (the median duration of hospitalization was 13.5 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic | Sugar Pill
Number analyzed (Participants) | 44 | 44
Participants | 9 | 12

ADVERSE EVENTS:
Arm/Group | Probiotic | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No